CLINICAL TRIAL: NCT01438892
Title: Impact Of RA Therapy Compliance On Patient-Reported Outcomes
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921144
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; therapy compliance
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- tDMARDs Group: traditional DMARDs
  Interventions: Drug: tDMARDs
- Biologics group: Biologics used in RA
  Interventions: Drug: biodmards

INTERVENTIONS:
Drug: tDMARDs — Traditional DMARDs for RA
  Groups: tDMARDs Group
Drug: biodmards — Biologic DMARDs
  Groups: Biologics group

SUMMARY:
Several observational studies have evaluated the comparative treatment costs associated with each agent, particularly those within the anti-TNF class, but few have evaluated the impact of therapy compliance, persistence, treatment patterns on patient reported outcomes, healthcare utilization and costs, using a provider database. This study is designed to fill in this information gap.

DETAILED DESCRIPTION:
Cohort observational

ELIGIBILITY:
Inclusion Criteria:

* Adults with moderate to severe RA who are currently using a DMARD

Exclusion Criteria:

* Psoriatic Arthritis (PsA), Psoriasis (PsO), SSystemic Lupus Erythematosus (SLE), Non-Disease modifying anti-rheumatic disease (non-DMARD) use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with modertate to severe Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
HAQ | 12 months
36-Item Short-Form Health Survey (SF-36) | 12 months

SECONDARY OUTCOMES:
Compliance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921144&StudyName=Impact%20Of%20RA%20Therapy%20Compliance%20On%20Patient-Reported%20Outcomes